CLINICAL TRIAL: NCT02754115
Title: A Prospective Audit of Perioperative Parameters of Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (CRS-HIPEC)
Brief Title: An Audit of Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Sohan Lal Solanki, Assistant Professor, Department of Anesthesiology, Critical Care and Pain, Tata Memorial Centre
Other Study IDs: PN 1667
Record Dates: First submitted 2016-03-29; First posted 2016-04-28 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Ovarian Cancer; Peritoneal Disease
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms; Peritoneal Diseases | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Hyperthermic intraperitoneal chemotherapy — Perioperative data of all the patients posted for cytoreductive surgery and hyperthermic intraperitoneal chemotherapy will be collected prospectively

SUMMARY:
Peritoneal carcinomatosis is a common event in the natural history of colorectal and other digestive tract cancers. Cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) provides a promising therapeutic option for highly selected patients with peritoneal carcinomatosis arising from different malignancies such as colorectal cancer, gastric cancer, ovarian cancer, or peritoneal mesothelioma with improvement of both patient survival and quality of life. CRS, i.e., removal of all visible metastatic abdominal and pelvic disease with peritonectomy along with HIPEC (for 90 min at a temperature of 42º C) and/or early postoperative intraperitoneal chemotherapy (EPIC) in order to eradicate all microscopic metastasis.

CRS with HIPEC is a long and complex procedure with significant blood and fluid loss during debulking, hemodynamic, hematological, and metabolic alterations before and during the HIPEC phase, and even in the early postoperative period, with resultant significant morbidity and mortality. Despite that most of the reported patients are in American Society of Anesthesiologist class I and II, without significant comorbidities or systemic disorder; the morbidity and mortality ranges from 12 to 65% in these procedures, so a well coordinated team of anesthesiologist, surgeons and intensivist and other ancillary services can result in good outcome. This study will see the challenges faced by the team regarding the pathophysiological alterations during the CRS with HIPEC in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years
2. ASA Class I to III
3. Colorectal and gynecological oncology cases posted for CRS with HIPC.

Exclusion Criteria:

1. Age less than 18 and more than 70 years
2. ASA Class IV and above

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: American Society of Anesthesiologist class I, II and III patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Changes in invasive blood pressure in perioperative period | From start of surgery upto 48 hours after surgery
  Invasive blood pressure will be measured in radial artery in perioperative period and changes from baseline will be recorded in a graphical manner
Changes in body temperature in perioperative period | From start of surgery upto 48 hours after surgery
  Body temperature will be measured in degree centigrade by nasopharyngeal temperature probe in perioperative period and changes from baseline will be recorded in a graphical manner
Changes in cardiac output in perioperative period | From start of surgery upto 48 hours after surgery
  Cardiac output will be measured in perioperative period and changes from baseline will be recorded in a graphical manner
Changes in arterial blood gas in perioperative period | From start of surgery upto 48 hours after surgery
  Arterial blood gases will be measured in perioperative period and changes from baseline will be recorded in a graphical manner

SECONDARY OUTCOMES:
Length of stay in intensive care unit | Upto 30 days after surgery
  Length of stay will be measured in days from admission to discharge in intensive care unit
Mortality | Upto 30 days after surgery
  30 days mortality will be noted if death occurred within this period

CONTACTS AND LOCATIONS:
Overall Officials: Sohan L solanki, Principal Investigator — Tata Memorial Centre
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Solanki SL, Agarwal V, Ambulkar RP, Joshi MP, Chawathey S, Rudrappa SP, Bhandare M, Saklani AP. The Hemodynamic Management and Postoperative Outcomes After Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy: A Prospective Observational Study. Crit Care Res Pract. 2024 Dec 27;2024:8815211. doi: 10.1155/ccrp/8815211. eCollection 2024. PMID 39760061